CLINICAL TRIAL: NCT05071092
Title: Dietary Intervention to Improve Health of Cardiovascular Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Gelderse Vallei Hospital (Other); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Renate Winkels, Renate Winkels, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL73021.091.20
Record Dates: First submitted 2021-08-27; First posted 2021-10-07 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Vascular Diseases
Keywords: Intervention study; RCT; nutrition; dietary guidelines; dietitian; cardiovascular diseases; tertiary prevention; SMART Risk Score
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The nature of the intervention does not allow for blinding of the participants or researchers. After data collection, the database will be coded by an independent researcher to ensure that data analysis is conducted in a blinded way.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention will consist of personalized guidance from a dietician focussing on improving adherence to the Dutch dietary guidelines.
  Interventions: Behavioral: Dietary counselling
- Usual care group (No Intervention): The usual care group will not receive any special guidance regarding healthy nutrition, but will have access to their care team as usual.

INTERVENTIONS:
Behavioral: Dietary counselling — Participants assigned to the intervention group will receive coaching from a dietitian to improve adherence to the Dutch dietary guidelines. Several behavioral change techniques will be used.
  Arms: Intervention group

SUMMARY:
Voed je Beter is a randomized, multicenter, controlled trial to examine whether personalized guidance to increase adherence to the Dutch dietary guidelines, compared to usual care, improves health of cardiovascular patients who receive regular medical treatment.

DETAILED DESCRIPTION:
Voed je Beter is a randomized, multicenter, controlled trial to examine whether a personalized intervention to increase adherence to the Dutch dietary guidelines, compared to usual clinical care, improves health of cardiovascular patients on top of medical treatment.

Patients previously diagnosed with cardiovascular disease are randomized into two parallel groups: the intervention or the usual care group. The intervention consists of personalized guidance from a dietician focussing on improving adherence to the Dutch dietary guidelines during a period of six months. The control group receives usual clinical care.

At baseline, three months, six months, and 12 months measurements will be performed. Primary outcome data will be collected at 6 months. After 12 months, additional data will be collected to assess the prolonged effects of the intervention. The primary outcome of interest is the difference in SMART Risk Score between the intervention and usual care group from baseline till six months.

Secondary outcomes are differences in SMART Risk Score at three months and twelve months; systolic blood pressure, diastolic blood pressure and cardiovascular parameters; diet quality, salt intake, vitamin levels in blood; body weight and waist circumference; renal function; quality of life; sleep; self-efficacy; mental health and medication use. In addition, an economic evaluation is carried out.

ELIGIBILITY:
Inclusion Criteria:

* A previously diagnosed cardiovascular disease, including acute coronary disease syndrome, angina pectoris, coronary revascularization, TIA, stroke, symptomatic aortic iliofemoral atherosclerosis, aortic aneurysm, intermittent claudication or peripheral revascularization.
* Over 18 years of age

Exclusion Criteria:

* Uses medication for treatment of diabetes
* A known hereditary form of cardiovascular diseases
* Chronic kidney disease stage 4 or above (eGFR<30)
* Participation in another research study of which the outcomes may interfere with the current trial
* Not able to speak and understand the Dutch language
* Unable/unwilling to comply with the intervention
* Active treatment for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Second manifestations of arterial disease (SMART) Risk Score | baseline till six months
  Estimate for 10-year risk for recurrent vascular events (range 0-100%), higher scores mean a worse outcome

SECONDARY OUTCOMES:
Second manifestations of arterial disease (SMART) Risk Score | baseline till three months, baseline till twelve months
  Estimate for 10-year risk for recurrent vascular events (range 0-100%), higher scores mean a worse outcome
Systolic and diastolic blood pressure | baseline, three months, six months and twelve months
  Blood pressure measurements following the recommendations for home blood pressure measurement by the European Society of Hypertension, meaning duplicate morning and evening measurements for 7 days.
Diabetic parameters | baseline, three months, six months and twelve months
  Insulin and glucose in mmol/L
Cardiovascular parameters | baseline, three months, six months and twelve months
  Total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides in mmol/L
Inflammation marker | baseline, three months, six months and twelve months
  HsCRP mg/l
Diet quality assessed by the Dutch Helathy Diet Index 2015 score (Eetscore-FFQ) | baseline, three months, six months and twelve months
  Dutch Healthy Diet Index 2015 score (range 0-160 points, higher scores mean better outcome), assessed by a short Food Frequency Questionnaire.
Salt intake | baseline, six months
  24-hour urinary sodium excretions.
Vitamin status | baseline, six months
  Serum vitamin B6, B12, folate and vitamin D.
Renal function | baseline, three months, six months and twelve months
  eGFR and albumin/creatinine ratio.
Anthropometrics - body weight | baseline, three months, six months and twelve months
  Body weight (in kilograms; weight and height will be combined to report BMI in kg/m^2)
Anthropometric - body height | baseline, three months, six months and twelve months
  Height (in meters; weight and height will be combined to report BMI in kg/m^2)
Anthropometrics -waist circumference | baseline, three months, six months and twelve months
  Waist circumference (in centimeters)
Self-reported quality of life | baseline, three months, six months and twelve months
  36-Item Short Form Health Survey questionnaire, a high score defines a more favorable health state.
Self-efficacy assessed by the Dutch general self-efficacy scale | baseline, three months, six months and twelve months
  Dutch general self-efficacy scale (range 10-40), a higher scores mean a more positive self-efficacy
Mental status: self-rating happiness | baseline, three months, six months and twelve months
  Single-item on a 7-point Likert scale
Mental status: self rated health | baseline, three months, six months and twelve months
  Single- item on a 5-point scale
Mental status: dispositional optimism | baseline, three months, six months and twelve months
  Life Orientation Test-Revised (LOT-R) 10-item questionnaire. The LOT-R sum score that ranges from 0 to 24, with higher scores indicating greater optimism.
Mental status: anxiety and depression symptoms | baseline, three months, six months and twelve months
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item depression module. The total score ranges from 0 to 27, with higher scores indicating higher severity of depressive symptoms
Mental status: depression symptoms | baseline, three months, six months and twelve months
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report screening scale with a score ranging from 0 to 21. Higher scores indicating higher severity of anxiety or depressive symptoms.
Evaluation from an economic perspective: quality of life | baseline, three months, six months and twelve months
  EuroQol- 5 Dimension questionnaire, the iMedical Consumption Questionnaire and the iProductivity Cost Questionnaire.
Evaluation from an economic perspective: productivity costs | baseline, three months, six months and twelve months
  The iProductivity Cost Questionnaire.
Evaluation from an economic perspective: medical consumption | baseline, three months, six months and twelve months
  The iMedical Consumption Questionnaire
Medication use | baseline, three months, six months and twelve months
  iMedical Consumption Questionnaire.
Sleep quality assessed by the Pittsburgh sleep quality index (PSQI) | baseline, three months, six months and twelve months
  The PSQI ranges from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Johanna M. Geleijnse, PhD, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] van Damme I, van Veldhuisen ER, Verkaar AJCF, Bemelmans RHH, Hovens MMC, Visseren FLJ, Koopal C, Winkels RM, Geleijnse JM. The effects of 6 months dietary counseling on diet quality and cardiovascular risk profile in patients with cardiovascular disease: A randomized controlled trial. Clin Nutr. 2025 Feb;45:101-110. doi: 10.1016/j.clnu.2024.12.020. Epub 2024 Dec 26. PMID 39798221

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT05071092/SAP_000.pdf